CLINICAL TRIAL: NCT00989053
Title: The Effect of SSRI Treatment on Affective Symptoms and Fertility Treatment Outcome in Women Undergoing In Vitro Fertilization for Unexplained Infertility - a Prospective Placebo-Controlled Study.
Brief Title: The Effect of Selective Serotonin Reuptake Inhibitor (SSRI) Treatment on Affective Symptoms and Fertility Treatment Outcome in Women Undergoing in Vitro Fertilization (IVF)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: dr.Gabi Aisenberg Romano M.D, Tel aviv Sourasky medical center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TASMC-09-GAR-078-CTIL
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2009-10-02 (Estimated); Status verified 2009-10

CONDITIONS: Depression; Anxiety; In Vitro Fertilization
Keywords: depression; anxiety; stress; antidepressant therapy; SSRI; infertility; in vitro fertilization (IVF); immunological factors; depressive and anxiety symptoms in women undergoing IVF treatment
MeSH Terms: conditions — Depression; Anxiety Disorders; Infertility | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- escitalopram (Active Comparator)
  Interventions: Drug: escitalopram; Drug: placebo
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: escitalopram — 10 mg/d for a duration of 8 weeks
  Arms: escitalopram
Drug: placebo — 1 pill per day for 8 weeks

SUMMARY:
Women undergoing IVF show a high prevalence of depressive and anxiety symptoms. Furthermore, stress has harmful consequences on IVF and pregnancy outcomes. An immunological cascade was suggested to be involved in the process. Treatment in this setting is usually psychotherapy rather than pharmacotherapy, despite reasonable biological evidence suggesting beneficial influence of antidepressant therapy on pregnancy and well-being. Moreover, pharmacotherapy is more available and affordable than psychotherapy in the public health system. The investigators suggest to study the efficacy of antidepressant treatment in women undergoing IVF treatment, presenting with mild mood symptoms. The investigators hypothesize that treatment will result in a greater attenuation of affective symptoms, as well as in higher pregnancy success rates. Furthermore, certain immunological stress-reactive factors, may prove to be the biological mechanism underlying these effects.

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 - 45 y.o.
2. A score higher then 45 on the Zung Self-Rating Anxiety Scale or a score higher then 16 on the Center for Epidemiologic Studies Depression Scale
3. Understanding of Hebrew
4. Willing to sign the informed consent

Exclusion Criteria:

1. An axis I DSM IVTR diagnosis other then a depressive, adjustment or anxiety disorder
2. Suicidal ideation
3. Current treatment with antidepressant medication
4. Physical illness explaining depressive symptoms (e.g. hypothyroidism, neurological disease, severe anemia, renal failure etc.)
5. Alcoholism or drug abuse and dependence
6. Past severe side effects to SSRIs
7. Failed IVF (4 trials of good quality embryo reinstatement without achieving pregnancy)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
positive blood βHCG | 2 months from date of signing informed consent

SECONDARY OUTCOMES:
psychiatric evaluation questionnaires | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel